CLINICAL TRIAL: NCT05608226
Title: Impact of Health Lifestyle on Body Weight Post Cessation of Pharmacotherapy in Obese Subjects
Brief Title: Impact of Health Lifestyle on Body Weight
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZSE-2210
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Body-Weight Trajectory
MeSH Terms: conditions — Body-Weight Trajectory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pharmacotherapy becomes an important and effective approach to improve body weight. However, it still remains unclear how to manage potential fluctuation after its cessation. Lifestyle change is the foundation and included as a part of clinical routine in real-world, therefore, we plan to conduct a prospective observational study to assess the impact of health lifestyle along with its compliance on body weight in Chinese people who live with obesity or overweight and are off-pharmacotherapy trial. The aim of this study is to examine the impact of health lifestyle along with its compliance on body weight related parameters in 6 months at 3 monthly intervals from treatment. In addition, body weight related results will be described.

DETAILED DESCRIPTION:
Novel pharmacotherapy is emerging, leading to substantial and sustained improvement in body weight compared with placebo in clinical trials. However, there is no evidence on management of body weight in real world setting after cessation of treatment. Body weight fluctuation is a pivotal difficulty for obese subjects who left off pharmacotherapy. It would be interesting to investigate the impact of real-world health lifestyle and its compliance in this clinical situation and probe into factors affecting compliance. Therefore, we will conduct a prospective observational study to assess the impact of health lifestyle along with its compliance on body weight in Chinese people who live with obesity or overweight and are off-pharmacotherapy trial. The aim of this study is to examine the impact of health lifestyle along with its compliance on body weight related parameters in 6 months at 3 monthly intervals from pharmacotherapy cessation. In addition, body weight related results will be described.

ELIGIBILITY:
Inclusion Criteria:

* All patients who completed a pharmacotherapy trial
* Those who consent to this FU study

Exclusion Criteria:

* Those who do not consent to this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who completed a pharmacotherapy trial will be recruited and who consent to this follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Fluctuation in body weight | 6 months
  To examine the weight fluctuation by health lifestyle compliance from baseline

SECONDARY OUTCOMES:
Change of blood lipids | 6 months
  To examine the change of blood lipids by health lifestyle compliance from baseline
Change of blood glucose levels | 6 months
  To examine the change of blood glucose levels by health lifestyle compliance from baseline
Change of blood pressure | 6 months
  To examine the change of blood pressure by health lifestyle compliance from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaoying Li, Shanghai, China

IPD SHARING:
Plan to Share IPD: No